CLINICAL TRIAL: NCT04197336
Title: Bariatric Embolization of Arteries With Imaging Visible Embolics
Brief Title: Bariatric Embolization of Arteries With Imaging Visible Embolics (BEATLES)
Acronym: BAE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00143169
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Morbid Obesity; Weight Loss
MeSH Terms: conditions — Obesity; Obesity, Morbid; Weight Loss

STUDY DESIGN:
Intervention Model Description: Pilot study
Masking Description: All participants in the pilot will receive study intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention (Experimental): There will be 10 pilot patients (See Statistical Analysis below for sample size calculations) for a total of 59 participants. Participants will be followed with study outcomes assessed for a period of 12 months. The duration of the study will be approximately three years.
  Interventions: Device: Bariatric Embolization of Arteries with imaging visible Embolics

INTERVENTIONS:
Device: Bariatric Embolization of Arteries with imaging visible Embolics — bariatric embolization will be performed using tiny (100-200 μm), radiopaque (visible on X-ray) beads (referred to as BTG-001933) in order to suppress the body's signals for feeling hungry, which we predict will lead to weight loss.
  Other Names: 100-200 µm radiopaque microspheres; Biocompatibles-001933

SUMMARY:
The BEATLES study is an investigator-initiated, prospective, double-blinded, randomized, sham-controlled study that will assess the impact of bariatric embolization on the systemic levels of obesity-related hormones and, as a consequence, on weight loss. The goal of this study is to help treat obesity combining a lifestyle program and a minimally invasive, angiographic (i.e., through blood vessels) approach.

DETAILED DESCRIPTION:
The BEATLES study is an investigator-initiated, prospective, double-blinded, randomized, sham-controlled study that will assess the impact of bariatric embolization on the systemic levels of obesity-related hormones and, as a consequence, on weight loss. The goal of this study is to help treat obesity combining a lifestyle program and a minimally invasive, angiographic (i.e., through blood vessels) approach.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥21 and ≤70 years
* Willing, able, and mentally competent to provide written informed consent
* Obese patients with a BMI ≥35 kg/m2
* Weight ≤400 lb
* Vascular anatomy (including celiac, hepatic, and gastric arteries) that in the opinion of the interventional radiologist is amendable to bariatric embolization, as assessed via 3D CT angiography
* Suitable for protocol therapy, as determined by the interventional radiology investigator
* Adequate hematologic (neutrophils>1.5x109/L, platelets>70x109/L, international normalized ratio (INR<1.5), hepatic (bilirubin≤2.0mg/dL, albumin≥2.5g/L), and renal (estimated glomerular filtration rate (GFR)>60milliliter mL/min. 1.73m2) function
* For females of reproductive potential: agreement to use of highly effective contraception
* for duration of study participation
* Patients who have failed conservative weight loss therapies such as supervised low calorie diets combined with behavior therapy and exercise
* Live or work within 65 miles of the enrolling institution in case a catastrophic post embolization event occurs

Exclusion Criteria:

* hemoglobin A1c greater than 8%
* Patients who are currently taking either Insulin or sulfonylurea (medication changes are allowed)
* Prior history of gastric, pancreatic, hepatic, and/or splenic surgery
* Prior radiation therapy to the upper abdomen
* Prior embolization to the stomach, spleen, or liver
* Cirrhosis
* Known portal venous hypertension
* Active peptic ulcer disease
* Significant risk factors for peptic ulcer disease, including daily NSAID use
* Large hiatal hernia, defined as >5 cm in size
* Active H. Pylori infection
* Known aortic pathology, such as aneurysm or dissection
* Renal insufficiency, as evidenced by an estimated glomerular filtration rate of <60 milliliter(mL)/min
* Major comorbidity, such as active cancer, significant cardiovascular disease, or peripheral arterial disease
* Pregnancy
* Pre-existing chronic abdominal pain
* Positive stool occult blood study
* GI bleeding or bleeding diathesis within 5 years
* Weight loss (intentional or unintentional) of more than or equal to 5% of body weight in the 6 months prior to randomization
* A weight loss greater than 6lb during the weight management run- in
* Use of anti-obesity medications in the 12 months prior to screening
* Endoscopic findings that would preclude bariatric embolization (at the discretion of the study team)
* History of gastric motility disorders or an abnormal nuclear gastric motility examination (to be performed in diabetic subjects only)
* American Society of Anesthesiologists Class 4 or 5 (very high risk surgical candidates: class 4=incapacitating disease that is a constant threat to life) at the time of screening for enrollment into the study - this exclusion criterion exists, because of the possibility that surgical intervention will be needed if the study intervention subsequently leads to severe adverse effects
* Inflammatory bowel disease
* Autoimmune disease or HIV+
* History of allergy to iodinated contrast media
* Failure to comply with pre-procedure weight management "run-in", or other pre-procedural visits (specifically, participants must complete 80% of weight management and Lose It! Food tracking, and 100% of one-time visits, i.e. MRI, computed tomography angiography (CTA), endoscopy)
* Applicability of any contraindication regarding patient's vasculature as per Instruction for Use
* Inability to have an MRI scan (i.e., metal implants or claustrophobia)
* Smokers/vape users/tobacco use
* Active or new-onset endocrine disorders (stable disease acceptable)
* Other unforeseen conditions that may make patients unsuitable for the procedure (study team discretion)

Exclusion Criteria (Psychiatric):

* As determined by clinical judgment based on Clinical Interview, psychological/behavioral measures, medical records, previous mental health records/other collateral information (as available) and consistent with diagnostic and statistical manual of mental disorders (DSM) -5 criteria:
* Diagnosis of severe mental illness (i.e., chronic psychotic spectrum disorders, clinically significant mood disorders) AND/OR one or more of the following:
* Evidence of active relapse or active impairing symptoms (e.g., suicidal ideation, audio or visual hallucinations, paranoia, thought disturbance, severe impairment)
* Evidence of minimal supports or limited adherence to ongoing mental health care
* Failure to provide comprehensive aftercare plan that includes emergency plan for addressing future mental health relapse
* History of treatment refractory mental illness/recurrent relapse (multiple suicide attempts or inpatient psychiatric hospitalizations in the past 5 years)
* Within past 3 years: Inpatient psychiatric hospitalization
* Within past 5 years: Suicide attempt
* Declining to provide mental health records, a letter of support from mental health professionals, or consent for verbal consultation with mental health professionals when determined to be essential to evaluation.
* Cognitive impairment, if judged to have
* Limited capacity to make informed decision about procedure and inability to verbalize an understanding of the surgical procedure, risks and benefits.
* Inability to demonstrate an understanding of the permanency of lifestyle change required
* History of Anorexia or History of/Active Bulimia: If determined to be of low enough severity not to be a clear contraindication, minimum of 5 years abstinence from bulimia, current moderate to severe binge eating or night eating syndrome
* Active or History of Substance Abuse with less than 5 years of abstinence
* Current use of anti-tricyclic anti-depressants or steroids, psychiatric medications associated with weight gain.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Weiss, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu Z, Cha SH, van Haasteren G, Wang J, Lane MD. Effect of centrally administered C75, a fatty acid synthase inhibitor, on ghrelin secretion and its downstream effects. Proc Natl Acad Sci U S A. 2005 Mar 15;102(11):3972-7. doi: 10.1073/pnas.0500619102. Epub 2005 Feb 23. PMID 15728730
- [Background] Loftus TM, Jaworsky DE, Frehywot GL, Townsend CA, Ronnett GV, Lane MD, Kuhajda FP. Reduced food intake and body weight in mice treated with fatty acid synthase inhibitors. Science. 2000 Jun 30;288(5475):2379-81. doi: 10.1126/science.288.5475.2379. PMID 10875926
- [Background] Cummings DE, Purnell JQ, Frayo RS, Schmidova K, Wisse BE, Weigle DS. A preprandial rise in plasma ghrelin levels suggests a role in meal initiation in humans. Diabetes. 2001 Aug;50(8):1714-9. doi: 10.2337/diabetes.50.8.1714. PMID 11473029
- [Result] Kojima M, Hosoda H, Date Y, Nakazato M, Matsuo H, Kangawa K. Ghrelin is a growth-hormone-releasing acylated peptide from stomach. Nature. 1999 Dec 9;402(6762):656-60. doi: 10.1038/45230. PMID 10604470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Ten pilot patients were enrolled. Due to funding, the study was stopped after 10 pilot patients.
Groups:
- Bariatric Embolization Procedure: Bariatric embolization will be performed using tiny (100-200 μm), radiopaque (visible on X-ray) beads (referred to as BTG-001933) in order to suppress the body's signals for feeling hungry.
Period: Overall Study
Arm/Group | Bariatric Embolization Procedure
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Bariatric Embolization Procedure: 10 subjects will be enrolled in the bariatric embolization(BM) pilot arm. BM procedure will be performed under moderate sedation. Procedure will take 1.5 hr to 3 hr subject will be placed on the X-ray fluoroscopy table. Radial or femoral vascular access will be achieved using a small gauge needle, dilated over a guidewire to accommodate a 5 French vascular sheath. Standard catheters, 3 dimensional imaging will be acquired of the stomach, the arteries supplying the fundus arising off the celiac vessel. Microcatheter into the left gastric and/or gastroepiploic arteries supplying the fundus and small calibrated spheres will be infused until stasis of anterograde arterial flow is achieved, with particular care to avoid infusion of non-target arteries. The left gastric and/or gastroepiploic arteries will be embolized. Repeat 3 dimensional imaging: assess bead distribution and fundal coverage. Subject will be monitored in the recovery room and will be observed overnight.
Arm/Group | Bariatric Embolization Procedure
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight as Assessed by BMI (kg/m^2)
Description: Efficacy of Bariatric Embolization procedure assessed by change in body weight as assessed by BMI.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Bariatric Embolization Procedure
Number analyzed (Participants) | 10
kg/m^2 | 43.7 (4.2)

2. Primary Outcome: Change in Body Weight (Pounds)
Description: Efficacy of Bariatric Embolization procedure assessed by change in body weight (pounds)
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Bariatric Embolization Procedure
Number analyzed (Participants) | 10
pounds | 14.3 (22.5)

ADVERSE EVENTS:
Time Frame: Up to 1 year
Groups:
- Pilot: Ten pilot participants will be used to test and refine the trial protocol, and data collection procedures.
Arm/Group | Pilot
All-Cause Mortality (participants affected / at risk) | 6/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilot (N=10)
Ucler (Gastrointestinal disorders) | 1 (1) — Deep gastric ulcer
Insomnia (General disorders) | 1 (1) — Insomnia
Site pseudoaneurysm (Vascular disorders) | 1 (1) — Embolization-unrelated vascular access site pseudoaneurysm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/36/NCT04197336/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT04197336/SAP_001.pdf
  • Informed Consent Form (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT04197336/ICF_002.pdf